CLINICAL TRIAL: NCT04806048
Title: Feasibility of the Use in Spanish Hospitals of Recommended Standards to Measure Results in Patients With Heart Failure (HF-Outcomes-Spain)
Brief Title: Feasibility of Implementation of Recommended Standards in Patients With Heart Failure
Acronym: HFOutcomesSP
Status: Completed | Type: Observational
Sponsor: Fundacion Profesor Novoa Santos (Other)
Collaborators: ODDS , S.L. (Unknown); Vifor Pharma España, S.L. (Unknown)
Responsible Party: Principal Investigator, Marisa Crespo Leiro, Head of Heart Failure Unit, Fundacion Profesor Novoa Santos
Other Study IDs: HF-Outcomes-Spain
Record Dates: First submitted 2020-12-22; First posted 2021-03-19 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
Keywords: Outcome; Heart-Failure; Standard of care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients and outpatients: There may be different types of patients with differing follow-up plan but all will bie considered one group regarding on whether they receive their recommended follow-up plan

SUMMARY:
Longitudinal pilot study among heart failure patients from six Spanish hospitals to evaluate the feasibility of establishing and maintaining for one year the set of standards for measuring results in patients with heart failure proposed by ICHOM (International Consortium for Health Outcomes Measurement), as well as identifying factors that hinder the use and applicability of this group of standards in real life, where appropriate, defined as the variables not filled in and the reason for the absence of such information.

DETAILED DESCRIPTION:
1. MAIN GOAL To evaluate through a pilot study the viability of establishing and maintaining for one year in selected Spanish centers the set of standards for measuring results in patients with heart failure proposed by ICHOM (International Consortium for Health Outcomes Measurement). (International Consortium for Health Outcomes Measurement).
2. SPECIFIC GOALS To identify factors that hinder the use and applicability of this group of standards in real life, where appropriate, defined as the variables not filled in and the reason for the absence of such information To estimate the workload necessary to implement this set of variables within everyday clinical practice.
3. STUDY DESIGN Observational pilot study with prospective follow-up with data collection at 30 days, 6 months and 1 year.

Due to the defined objective, the methods used are, to a large extent, those proposed by ICHOM, except in those sections that may be slightly modified to adapt to the local situation.

3.1. Selection of centers and patients Six centers with experience and adequate organization (heart failure unit) and with a sufficient size have been selected to guarantee the recruitment of patients in a short period of time (around three weeks). The main justification was to seek, within the usual clinical practice, centers where, due to the organization and interest in heart failure, the chances of success of this initiative were greater.

100 consecutive patients with a diagnosis of heart failure who meet inclusion criteria and with no exclusion criteria will be selected in each center.

3.2. Sample size considerations For the main outcome, success is considered if the proportion of patients followed is ≥ 70%. A random sample of 588 individuals is sufficient to estimate, with 95% confidence and a precision of +/- 3.5 percentage units, a population percentage that is expected to be around 75%. Six Spanish centers will participate and a recruitment target of 100 consecutive patients is set, for a total of 600 patients in the study. In addition, these sizes in each center offer, accepting an alpha risk of 0.05, a power greater than 80% to detect statistically significant differences between two centers, assuming that a follow-up of 75% of patients is achieved in one and 55% in the other.

3.3. Follow-up From the baseline or inclusion visit and afterwards, in newly diagnosed patients or in those recruited in an acute situation, follow-up visits at 30 days, 6 months and 1 year [Hospitalized patients (1. A recent diagnosis, that is, they did not previously have the diagnosis of HF and 2.Patients with a previous diagnosis of HF and who are admitted for an episode of decompensation of HF) and Outpatients (1. A recent diagnosis that is in the process of titration and/or compensation and 2.A previous diagnosis, that they have suffered a decompensation, either defined because they have had to go to the emergency room or have been seen in the outpatient clinic for that reason)].

In patients who were included in a stable situation, the 30-day visit will not be carried out (Outpatients: "Stable" patients attending a follow-up visit. A simple follow-up) since doing so would unjustifiably complicate the follow-up, giving more work and discomfort to patients and health professionals. The outcomes reported by the patient (PROMs) in the visits every six months may be collected by telephone contact if the doctor, due to the stable situation of the patient, does not consider the face-to-face visit necessary. Information will be collected at in the case of hospital admissions during follow-up, these admissions also set the "counter to zero" with regard to time for the following visits (30 days, six months…).

4. DATA COLLECTION AND MANAGEMENT A data entry application will be enabled that will include filters to detect inconsistencies and anomalous data and alarms for patient monitoring. The data will be anonymized for all the people involved in the study except for the person in charge in each center, who will be able to identify their patients to enable follow-up.

5. PLAN FOR DATA ANALYSIS Two data analyses are planned, one that includes the information from the baseline visit and the 30-day visit (in patients for whom it is indicated in the protocol) and the final one with all the information collected. In both cases, a global analysis and a comparison between centers (benchmarking) will be carried out.

In line with the main objective of this pilot study, the main variables are the proportion of patients who remain in follow-up, the proportion of patients in whom follow-up is carried out, in terms of time, as planned, and the proportion of missing data in each one of the defined outcomes.

The pilot's success criteria will be a follow-up> 70%, a proportion of missing data in the outcomes <10%.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Diagnosed with heart failure: Clinical identification of signs and symptoms of heart failure and objective evidence of heart dysfunction.
* Acute presentation (first presentation or decompensation of already known HF, whether or not it causes hospital admission) or chronic (stable outpatients) of any etiology
* Any value of the ejection fraction.
* Give writed informed consent to participate in the study.

Exclusion Criteria:

* Patients whose first manifestation of heart failure is cardiogenic shock, in that first episode. Those patients who survived an initial episode of shock and remain in heart failure can be included once stabilized.
* Heart transplant patients
* Patients with long-lasting ventricular assist devices
* Patients with isolated right heart failure.
* Patients with onset of heart failure and whose cause can be corrected immediately (eg, acute ischemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the situation at the time of inclusion,5 types of patients are defined that reflect different clinical situations and influence the necessary follow-up plan.
  A.Hospitalized patients:
  1. A recent diagnosis (at that admission), that is, they did not previously have the diagnosis of HF
  2. Patients with a previous diagnosis of HF and who are admitted for an episode of decompensation of HF.
  B.Outpatients:
  1. A recent diagnosis that is in the process of titling and/or compensation
  2. A previous diagnosis, that they have suffered a decompensation, well defined because they have had to go to the emergency room (and the diuretic treatment has been increased) or have been seen in the outpatient clinic for that reason
  3. "Stable" patients attending a follow-up visit.A simple follow-up
Sampling Method: Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Patients in follow-up | Up to 1 year
  Proportion of patients who receive their recommended follow-up plan

CONTACTS AND LOCATIONS:
Overall Officials: María G Crespo Leiro, MD, Principal Investigator — Complejo Hospitalario Universitario de A Coruña (CHUAC)
Locations (6):
- Spain (6):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groenewegen A, Rutten FH, Mosterd A, Hoes AW. Epidemiology of heart failure. Eur J Heart Fail. 2020 Aug;22(8):1342-1356. doi: 10.1002/ejhf.1858. Epub 2020 Jun 1. PMID 32483830
- [Background] Anguita Sanchez M, Crespo Leiro MG, de Teresa Galvan E, Jimenez Navarro M, Alonso-Pulpon L, Muniz Garcia J; PRICE Study Investigators. Prevalence of heart failure in the Spanish general population aged over 45 years. The PRICE Study. Rev Esp Cardiol. 2008 Oct;61(10):1041-9. doi: 10.1016/s1885-5857(09)60007-4. PMID 18817680
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] Anguita Sanchez M, Lambert Rodriguez JL, Bover Freire R, Comin Colet J, Crespo Leiro MG, Gonzalez Vilchez F, Manito Lorite N, Segovia Cubero J, Ruiz Mateas F, Elola Somoza FJ, Iniguez Romo A. Classification and Quality Standards of Heart Failure Units: Scientific Consensus of the Spanish Society of Cardiology. Rev Esp Cardiol (Engl Ed). 2016 Oct;69(10):940-950. doi: 10.1016/j.rec.2016.06.006. Epub 2016 Aug 27. English, Spanish. PMID 27576081
- [Background] McDonagh TA, Blue L, Clark AL, Dahlstrom U, Ekman I, Lainscak M, McDonald K, Ryder M, Stromberg A, Jaarsma T; European Society of Cardiology Heart Failure Association Committee on Patient Care. European Society of Cardiology Heart Failure Association Standards for delivering heart failure care. Eur J Heart Fail. 2011 Mar;13(3):235-41. doi: 10.1093/eurjhf/hfq221. Epub 2010 Dec 15. PMID 21159794
- [Background] Burns DJP, Arora J, Okunade O, Beltrame JF, Bernardez-Pereira S, Crespo-Leiro MG, Filippatos GS, Hardman S, Hoes AW, Hutchison S, Jessup M, Kinsella T, Knapton M, Lam CSP, Masoudi FA, McIntyre H, Mindham R, Morgan L, Otterspoor L, Parker V, Persson HE, Pinnock C, Reid CM, Riley J, Stevenson LW, McDonagh TA. International Consortium for Health Outcomes Measurement (ICHOM): Standardized Patient-Centered Outcomes Measurement Set for Heart Failure Patients. JACC Heart Fail. 2020 Mar;8(3):212-222. doi: 10.1016/j.jchf.2019.09.007. Epub 2019 Dec 11. PMID 31838032
- [Background] McNamara RL, Spatz ES, Kelley TA, Stowell CJ, Beltrame J, Heidenreich P, Tresserras R, Jernberg T, Chua T, Morgan L, Panigrahi B, Rosas Ruiz A, Rumsfeld JS, Sadwin L, Schoeberl M, Shahian D, Weston C, Yeh R, Lewin J. Standardized Outcome Measurement for Patients With Coronary Artery Disease: Consensus From the International Consortium for Health Outcomes Measurement (ICHOM). J Am Heart Assoc. 2015 May 19;4(5):e001767. doi: 10.1161/JAHA.115.001767. PMID 25991011

DOCUMENTS (1):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT04806048/Prot_000.pdf